CLINICAL TRIAL: NCT03008967
Title: A Prospective Cohort Study of Patients Undergoing Total Knee and Hip Arthroplasty at a Regional Hospital in Denmark
Brief Title: A Study of Patients Undergoing Total Knee and Hip Arthroplasty at a Regional Hospital in Denmark
Status: Completed | Type: Observational
Sponsor: Bornholms Regionskommune (Other Government)
Responsible Party: Principal Investigator, Troels Mark Christensen, Physiotherapist, B.Pt., M.Sc., Bornholms Regionskommune
Other Study IDs: 2016-41-4783
Record Dates: First submitted 2016-09-09; First posted 2017-01-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Arthroplasty, Replacement, Knee; Arthroplasty, Replacement, Hip
Keywords: Total Knee Arthroplasty; Total Hip Arthroplasty; Rehabilitation
MeSH Terms: interventions — Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Knee and Hip Arthroplasty: Rehabilitation, observational. Identification of risk factors for poor response to rehabilitation programs after TJR and use these to identify patients who are most susceptible to poor outcomes
  Interventions: Other: Arthroplasty and postoperative rehabilitation.

INTERVENTIONS:
Other: Arthroplasty and postoperative rehabilitation. — Patients undergoing total knee or total hip arthroplasty and their response to postoperative rehabilitation.

SUMMARY:
This project will be a descriptive, hypothesis-generating study. The aim is to identify risk factors for poor response to rehabilitation programs after TJR and use these to identify patients who are most susceptible to poor outcomes in order to optimise appropriate rehabilitations strategies and rationalising the distribution of health care resources.

DETAILED DESCRIPTION:
Fast-track surgery for total knee and hip arthroplasty has improved markedly in recent years with decreased hospitalization and postoperative complications. In 2014 there were performed over 9000 total hip arthroplasty (THA) and over 8500 total knee arthroplasty operations (TKA) in Denmark. During the same year Bornholm's regional hospital performed 85 THA's and 47 TKA's of these operations.

Even though the initial surgical procedure being technical and radiological satisfactory, there are a big proportion of patients who endure dissatisfaction and disability after total joint replacement (TJR) (between 20-40%). The strongest predictor for dissatisfaction after a TKA were found to be preoperative expectation not met postoperatively (10.7x greater risk). To date, there is no criterion standard for assessing the outcome of neither expectations nor satisfaction for patients undergoing TJR.

Patient's expectations are of a particular significance because they are linked to requests for elective and often costly treatments. Several studies have investigated the fulfillment of patient' expectations, however the focus has been primarily assessed by expectations regarding pain, but may also be influenced by several other factors. Patient's expectations are also strongly related to patient's assessments of outcome.

It is well established that there is a correlation between satisfaction of surgery and objective improvements in pain, function and general health-related quality of life, but just as patient' expectations the postoperative satisfaction may also incorporate multiple and varies factors that affect the overall outcome. One of these factors can be "ability to forget the artificial joint" in everyday life and can therefore be regarded as the ultimate possible goal for patient satisfaction.

Additionally, many patients undergoing TJR experience continued disability, which is largely caused by persistent pain postoperatively. Studies have shown that a high level of pain catastrophizing is a predictor of high levels of acute and persistent pain after various surgeries, and further investigation of pain catastrophizing as a predictor of outcome after TJR is warranted.

Many of the patients who experience dissatisfaction and disability after TJR do not undergo revision and present a burden for the community health clinicians and health services to continue to remedy their dissatisfaction. The rehabilitation after the initial surgery has been proven to produce short-term benefits, but these benefits does not seem to persist. As many patients' experiences limited clinical improvements postoperatively and no national consensus on the rehabilitation for this group, an optimal rehabilitation protocol for this group of patients is still warranted.

Several other associations between patient characteristics and the chance to achieve clinically importance improvements to TJR surgery have been identified as age, gender, body mass index, ethnicity, psychological distress, co-morbidity-profile and radiographic osteoarthritis severity. It can be speculated that while fast-track surgery aid to early recovery, the number of falls within the population of patients undergoing total lower limb arthroplasty will increase as a result from increased, early activities. Jørgensen & Kehlet found the overall incidence of falls postoperatively in hip and knee replacements to be low, the inclusion of fall history may be important to optimize the rehabilitation protocol and reduce future risk of falls in this group of patients.

Patients undergoing lower TJR wish to return to pre-pathological physical status, but there has been found a limited interest in actually undertaking greater efforts in physical therapy to fully achieve this either for pleasure or health gains. Individual beliefs and perceptions presents a big factor influencing physical activity postoperatively and it is therefore important to examine this further when developing management plans aimed to optimize rehabilitation in this group of patients.

There is a dearth of literature examining the impact on actual response rates in rehabilitation after TJR surgery taken fall history, patient expectations, subjective as well as objective measurements into account. It is therefore important to clarify the relationship between these characteristics and responsiveness to postoperative rehabilitation. The available data suggest that identifying and addressing the mechanism for reduced activity and identification of the group of patients who may or may not benefit from a rehabilitation programme may be the approach needed. This data can be used to allocate already sparse resources more beneficially, and to optimise criteria for the rehabilitation intervention. An expert consensus on the best practice has already identified the need for preoperative screening to identify patients most in need for rehabilitation for patients undergoing total hip arthroplasty.

Aim:

This project will be a descriptive, hypothesis-generating study. The aim is to identify risk factors for poor response to rehabilitation programs after TJR and use these to identify patients who are most susceptible to poor outcomes in order to optimise appropriate rehabilitations strategies and rationalising the distribution of health care resources.

Material and methods:

This project will be of a prospective cohort design where all patients who are scheduled to undergo a total joint replacement (total knee arthroplasty or total hip arthroplasty) at Bornholms regional hospital will be invited to participate. Due to the minimal effort and time required filling out the questionnaires and performing the 30sec chair stand test a minimal number of patients are expected to decline participation. Based on clinical experience the annual number of patients to undergo lower extremity TJR at Bornholm's regional hospital is expected to be around 160 patients.

During study enrolment basic, demographic data (e.g. age, gender, co-morbidities, BMI) will be collected on each participant.

Preoperative assessments (prior to surgery) and postoperative assessments (follow up at 3 months after surgery) will include:

Preoperative assessments:

* Use of joint specific analgesics and other medication
* Fall history
* Patient expectation questionnaire
* Pain catastrophizing questionnaire
* KOOS / HOOS questionnaire
* 30 second chair stand test

Postoperative assessments:

* Use of joint specific analgesics and other medication
* Fall history
* KOOS / HOOS questionnaire
* Pain catastrophizing questionnaire
* 30 second chair stand test
* The Forgotten Joint Score
* Patient satisfaction questionnaire

Approvals:

This cohort study has to obtain approval from the Danish Datatilsynet (J.nr. 2016-41-4783). This study will not change the pre or postoperative treatment of the included patients, and therefore no other formal approval is required.

Postoperative rehabilitation:

All patients are given a rehabilitation plan from the hospital to engage in a 4-12 weeks rehabilitation program in one of two rehabilitations centres located on Bornholm. The rehabilitation starts with a individual consultation with an experienced physiotherapist within 3 weeks of surgery where appropriate home-exercises are revised and instructed, and shortly after the consultation the patient is enrolled in a out-patient, group-based physical therapy program, twice weekly sessions for 4-12 weeks, where the length of the program depends on the patients objective response to the physical therapy. The patients are encouraged to continue their home-based exercises parallel to the physical therapy sessions and after the culmination of the physical therapy program. At the end of the supervised physical therapy program, the involved physiotherapist will subjectively assess each patient's compliance in regards to their exercise adherence to the rehabilitation the patients have undertaken.

Evaluation of the surgery and rehabilitation intervention is performed at the hospital 3 months after the surgery by the assigned orthopaedic surgeon, where the postoperatively outcome measurements will be recorded.

Statistical analysis:

The statistical analysis will compare preoperative and postoperative scores in terms of the use of analgesics, fall history, patient expectations / satisfaction, KOOS / HOOS, pain catastrophizing, the forgotten joint score and 30sec chair stand test. Significance will be set to <0.05. A Chi-square test will be used to investigate whether distributions of categorical variables differ from one another. Multivariable linear regression will be performed to examine the association between patient characteristics and the response rate to TKA and THA individually and TKA/THA combined.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing total knee arthroplasty or total hip arthroplasty
* must be able to participate in postoperative rehabilitation
* must be able to talk and understand Danish or English

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are scheduled to undergo a total joint replacement (total knee arthroplasty or total hip arthroplasty) at Bornholms regional hospital will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
30 second chair stand test, to test the patients functional capacity | Change of 30 second chair stand test from baseline to follow up (an average of 3 months)

SECONDARY OUTCOMES:
Health-related quality of life questionnaire | Change of health-related quality of life questionnaire from baseline to follow up (an average of 3 months)
  Knee injury and Osteoarthritis Outcome Score (KOOS) or Hip disability and Osteoarthritis Outcome Score (HOOS)
Pain catastrophizing scale questionnaire | Change of pain catastrophizing scale questionnaire from baseline to follow up (an average of 3 months)
Use of analgesics and other medication, qualitative assessment | Changes in the use og analgesics and other medication from baseline to follow up (an average of 3 months)
Fall history, events as numbers of falls described by the patient | Change within the fall history from baseline to follow up (an average of 3 months)
Patient expectations questionnaire | Preoperative (an average 3 weeks before surgery)
Patient satisfaction questionnaire | At follow up (an average of 3 months postoperative).
The Forgotten Joint Score questionnaire | At follow up (an average of 3 months postoperative).
Rehabilitation compliance | At the culmination of the rehabilitation program, an average of 10 weeks.
  Physiotherapist subjective assessment of patient compliance to the rehabilitation program

CONTACTS AND LOCATIONS:
Overall Officials: Troels M. Christensen, MSc, Principal Investigator — Bornholms Regionskommune
Locations (1):
- Genoptræningen, Rønne, Bornholm, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Aasvang EK, Luna IE, Kehlet H. Challenges in postdischarge function and recovery: the case of fast-track hip and knee arthroplasty. Br J Anaesth. 2015 Dec;115(6):861-6. doi: 10.1093/bja/aev257. Epub 2015 Jul 25. PMID 26209853
- [Background] Artz N, Elvers KT, Lowe CM, Sackley C, Jepson P, Beswick AD. Effectiveness of physiotherapy exercise following total knee replacement: systematic review and meta-analysis. BMC Musculoskelet Disord. 2015 Feb 7;16:15. doi: 10.1186/s12891-015-0469-6. PMID 25886975
- [Background] Behrend H, Giesinger K, Giesinger JM, Kuster MS. The "forgotten joint" as the ultimate goal in joint arthroplasty: validation of a new patient-reported outcome measure. J Arthroplasty. 2012 Mar;27(3):430-436.e1. doi: 10.1016/j.arth.2011.06.035. Epub 2011 Oct 13. PMID 22000572
- [Background] Bourne RB, Chesworth BM, Davis AM, Mahomed NN, Charron KD. Patient satisfaction after total knee arthroplasty: who is satisfied and who is not? Clin Orthop Relat Res. 2010 Jan;468(1):57-63. doi: 10.1007/s11999-009-1119-9. PMID 19844772
- [Background] Burns LC, Ritvo SE, Ferguson MK, Clarke H, Seltzer Z, Katz J. Pain catastrophizing as a risk factor for chronic pain after total knee arthroplasty: a systematic review. J Pain Res. 2015 Jan 5;8:21-32. doi: 10.2147/JPR.S64730. eCollection 2015. PMID 25609995
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Di Monaco M, Castiglioni C. Which type of exercise therapy is effective after hip arthroplasty? A systematic review of randomized controlled trials. Eur J Phys Rehabil Med. 2013 Dec;49(6):893-907, quiz 921-3. Epub 2013 Oct 30. PMID 24172644
- [Background] Dobson F, Hinman RS, Hall M, Terwee CB, Roos EM, Bennell KL. Measurement properties of performance-based measures to assess physical function in hip and knee osteoarthritis: a systematic review. Osteoarthritis Cartilage. 2012 Dec;20(12):1548-62. doi: 10.1016/j.joca.2012.08.015. Epub 2012 Aug 31. PMID 22944525
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Dowsey MM, Gunn J, Choong PF. Selecting those to refer for joint replacement: who will likely benefit and who will not? Best Pract Res Clin Rheumatol. 2014 Feb;28(1):157-71. doi: 10.1016/j.berh.2014.01.005. PMID 24792950
- [Background] Granot M, Ferber SG. The roles of pain catastrophizing and anxiety in the prediction of postoperative pain intensity: a prospective study. Clin J Pain. 2005 Sep-Oct;21(5):439-45. doi: 10.1097/01.ajp.0000135236.12705.2d. PMID 16093750
- [Background] Harding PA, Holland AE, Hinman RS, Delany C. Physical activity perceptions and beliefs following total hip and knee arthroplasty: a qualitative study. Physiother Theory Pract. 2015 Feb;31(2):107-13. doi: 10.3109/09593985.2014.959581. Epub 2014 Dec 12. PMID 25495877
- [Background] Jorgensen CC, Kehlet H; Lundbeck Foundation Centre for Fast-track Hip and Knee Replacement Collaborative Group. Fall-related admissions after fast-track total hip and knee arthroplasty - cause of concern or consequence of success? Clin Interv Aging. 2013;8:1569-77. doi: 10.2147/CIA.S52528. Epub 2013 Nov 26. PMID 24348026
- [Background] Kehlet H. Fast-track hip and knee arthroplasty. Lancet. 2013 May 11;381(9878):1600-2. doi: 10.1016/S0140-6736(13)61003-X. No abstract available. PMID 23663938
- [Background] Kjogx H, Zachariae R, Pfeiffer-Jensen M, Kasch H, Svensson P, Jensen TS, Vase L. Pain frequency moderates the relationship between pain catastrophizing and pain. Front Psychol. 2014 Dec 19;5:1421. doi: 10.3389/fpsyg.2014.01421. eCollection 2014. PMID 25646089
- [Background] Lynge E, Sandegaard JL, Rebolj M. The Danish National Patient Register. Scand J Public Health. 2011 Jul;39(7 Suppl):30-3. doi: 10.1177/1403494811401482. PMID 21775347
- [Background] Mancuso CA, Jout J, Salvati EA, Sculco TP. Fulfillment of patients' expectations for total hip arthroplasty. J Bone Joint Surg Am. 2009 Sep;91(9):2073-8. doi: 10.2106/JBJS.H.01802. PMID 19723982
- [Background] Mancuso CA, Salvati EA, Johanson NA, Peterson MG, Charlson ME. Patients' expectations and satisfaction with total hip arthroplasty. J Arthroplasty. 1997 Jun;12(4):387-96. doi: 10.1016/s0883-5403(97)90194-7. PMID 9195314
- [Background] Mancuso CA, Sculco TP, Salvati EA. Patients with poor preoperative functional status have high expectations of total hip arthroplasty. J Arthroplasty. 2003 Oct;18(7):872-8. doi: 10.1016/s0883-5403(03)00276-6. PMID 14566742
- [Background] Mancuso CA, Sculco TP, Wickiewicz TL, Jones EC, Robbins L, Warren RF, Williams-Russo P. Patients' expectations of knee surgery. J Bone Joint Surg Am. 2001 Jul;83(7):1005-12. doi: 10.2106/00004623-200107000-00005. PMID 11451969
- [Background] Nilsdotter A, Bremander A. Measures of hip function and symptoms: Harris Hip Score (HHS), Hip Disability and Osteoarthritis Outcome Score (HOOS), Oxford Hip Score (OHS), Lequesne Index of Severity for Osteoarthritis of the Hip (LISOH), and American Academy of Orthopedic Surgeons (AAOS) Hip and Knee Questionnaire. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S200-7. doi: 10.1002/acr.20549. No abstract available. PMID 22588745
- [Background] Nilsdotter AK, Lohmander LS, Klassbo M, Roos EM. Hip disability and osteoarthritis outcome score (HOOS)--validity and responsiveness in total hip replacement. BMC Musculoskelet Disord. 2003 May 30;4:10. doi: 10.1186/1471-2474-4-10. Epub 2003 May 30. PMID 12777182
- [Background] Nilsdotter AK, Toksvig-Larsen S, Roos EM. Knee arthroplasty: are patients' expectations fulfilled? A prospective study of pain and function in 102 patients with 5-year follow-up. Acta Orthop. 2009 Feb;80(1):55-61. doi: 10.1080/17453670902805007. PMID 19234886
- [Background] Palazzo C, Jourdan C, Descamps S, Nizard R, Hamadouche M, Anract P, Boisgard S, Galvin M, Ravaud P, Poiraudeau S. Determinants of satisfaction 1 year after total hip arthroplasty: the role of expectations fulfilment. BMC Musculoskelet Disord. 2014 Feb 24;15:53. doi: 10.1186/1471-2474-15-53. PMID 24564856
- [Background] Pavlin DJ, Sullivan MJ, Freund PR, Roesen K. Catastrophizing: a risk factor for postsurgical pain. Clin J Pain. 2005 Jan-Feb;21(1):83-90. doi: 10.1097/00002508-200501000-00010. PMID 15599135
- [Background] Rolfson O, Bohm E, Franklin P, Lyman S, Denissen G, Dawson J, Dunn J, Eresian Chenok K, Dunbar M, Overgaard S, Garellick G, Lubbeke A; Patient-Reported Outcome Measures Working Group of the International Society of Arthroplasty Registries. Patient-reported outcome measures in arthroplasty registries Report of the Patient-Reported Outcome Measures Working Group of the International Society of Arthroplasty Registries Part II. Recommendations for selection, administration, and analysis. Acta Orthop. 2016 Jul;87 Suppl 1(Suppl 1):9-23. doi: 10.1080/17453674.2016.1181816. Epub 2016 May 26. PMID 27228230
- [Background] Roos EM, Roos HP, Lohmander LS, Ekdahl C, Beynnon BD. Knee Injury and Osteoarthritis Outcome Score (KOOS)--development of a self-administered outcome measure. J Orthop Sports Phys Ther. 1998 Aug;28(2):88-96. doi: 10.2519/jospt.1998.28.2.88. PMID 9699158
- [Background] Smith TO, Latham S, Maskrey V, Blyth A. Patients' perceptions of physical activity before and after joint replacement: a systematic review with meta-ethnographic analysis. Postgrad Med J. 2015 Sep;91(1079):483-91. doi: 10.1136/postgradmedj-2015-133507. Epub 2015 Aug 25. PMID 26306502
- [Background] Thomsen MG, Latifi R, Kallemose T, Barfod KW, Husted H, Troelsen A. Good validity and reliability of the forgotten joint score in evaluating the outcome of total knee arthroplasty. Acta Orthop. 2016 Jun;87(3):280-5. doi: 10.3109/17453674.2016.1156934. Epub 2016 Mar 3. PMID 26937689
- [Background] Westby MD, Brittain A, Backman CL. Expert consensus on best practices for post-acute rehabilitation after total hip and knee arthroplasty: a Canada and United States Delphi study. Arthritis Care Res (Hoboken). 2014 Mar;66(3):411-23. doi: 10.1002/acr.22164. PMID 24023047
- [Background] Thomsen, M. G. (2015). Comparison of Vanguard XP and Vanguard CR Total Knee Arthroplasties. A Trial Evaluating Early Component Migration by RSA and Patient Reported Outcome. Study is ongoing.